CLINICAL TRIAL: NCT00527982
Title: Celecoxib as Adjuvant Biologic Therapy in Patients With Early Stage Head and Neck and Lung Cancer
Brief Title: Celecoxib as Adjuvant Biologic Therapy in Patients With Head and Neck and Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Termination due to poor accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0104
Record Dates: First submitted 2007-09-10; First posted 2007-09-11 (Estimated); Results first posted 2011-04-20 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Head and Neck Cancer; Lung Cancer
Keywords: Head and Neck Cancer; Lung Cancer; Non-Small Cell Lung Cancer; Celecoxib; Celebrex
MeSH Terms: conditions — Head and Neck Neoplasms; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Celecoxib treatment (Experimental): 600 mg orally (PO) daily
  Interventions: Drug: Celecoxib
- No treatment (No Intervention)

INTERVENTIONS:
Drug: Celecoxib — 600 mg by mouth daily for a total of 12 months.
  Other Names: Celebrex
  Arms: Celecoxib treatment

SUMMARY:
Primary Objectives:

1. To examine the effect of celecoxib treatment on histological response, markers of proliferation (Ki-67), and apoptosis. Secondary endpoints include time to second primary or recurrence and survival.
2. To examine the toxicity associated with celecoxib administration in patients with previously treated Head and Neck Head and neck squamous cell carcinomas (HNSCC)or Non-small-cell lung carcinoma (NSCLC).

DETAILED DESCRIPTION:
In order to enroll in this trial, you must also be enrolled in Protocol 2003-0424. The study procedures and tests that are part of this study are the same procedures and tests that are part of Protocol 2003-0424. Even though a procedure or test is described in both this consent and the consent for Protocol 2003-0424, you will only have the described procedure or test done once. For example, both this study and Protocol 2003-0424 require a complete physical exam before beginning treatment. In this case, you will only have one physical exam that will count for both studies.

Celecoxib is a drug that slows the production of chemicals in the body that cause inflammation. Celecoxib works by interfering with the action of the chemical cyclooxygenase, a chemical that is involved in inflammation. It is believed that the product of chemicals that cause inflammation may be involved in cancer development.

Before treatment starts, you will have a complete physical exam, including measurement of height, weight, blood pressure, and vital signs. You will have blood samples drawn for routine blood tests (about 3 teaspoons) and for research purposes (about 4 teaspoons) . Women who are able to have children must have a negative pregnancy test (blood or urine). You will also have a chest x-ray and a CT scan of your chest.

You will also have a bronchoscopy (tissue sample from the lung) at the beginning of this study for lab analysis. For this procedure, you will be given drugs to relax. Then, a local anesthetic will be sprayed in your nose and throat to numb those areas. A slim, flexible tube with a light will be placed through your nose or mouth and into your lungs. Tweezers will be fed through the tube to collect lung tissue (biopsy) samples from 6 different places in your lungs. During the bronchoscopy procedure, a complete inspection of the airways will be performed. Any suspicious areas that are seen under the white-light and autofluorescence bronchoscopy will be identified and more biopsies and brushings will be performed to evaluate whether any pre-cancerous tissue is present. You will also have a bronchial brushing next to each biopsy site. In a bronchial brushing, a small brush is fed through the tube into your lungs and a sample of lung tissue is gently scraped off. When the biopsies and brushings are done, you will have a bronchial lavage (bronchial washing). In the bronchial lavage, a small amount of water (about 4 tablespoons) is sprayed into your lungs and then suctioned out through the tube. This fluid is used to collect additional tissue and mucous samples. In addition, a sputum (saliva) sample will be taken and the inside of your cheek will be scraped (buccal sample).

If you have had HNSCC, you will also have a laryngoscopy. In a laryngoscopy, a lighted tube is placed down your throat and the larynx is checked. The back of your throat will be sprayed with an anesthetic before this procedure to make the procedure more comfortable.

In this study you will be randomly assigned (as in the toss of a coin) to one of two groups. Participants in one group will receive celecoxib. Participants in the other group will receive no treatment. Current standard practice for individuals who have had therapy for early stage NSCLC or HNSCC is follow-up (no treatment). You have a 2 to 1 chance of being assigned to the treatment group. That means that 2 out of every 3 participants in this study will be assigned to the treatment group.

If you are assigned to the treatment group you will take celecoxib by mouth in two divided doses at least 8 hours apart every day. Your study doctor will tell you exactly how many pills you should take each day. You will take celecoxib for up to 12 months. You will be taken off study if intolerable side effects occur or if the disease comes back.

If you are assigned to the treatment (celecoxib) group, you will have a physical exam by a physician or nurse at months 3, 6, and 12 for the first year of treatment. If you are assigned to the "no treatment" group, the nurse will contact you by phone every 3 months for the first year on this study to see how you are doing and you will have a physical exam by either a physician or a nurse every 6 months. During the first year, all participants will have blood samples taken at each clinic visit for routine blood tests (about 3 teaspoons) and for research purposes (about 4 teaspoons). In addition, all participants will have a chest x-ray and chest CT at months 6 and 12. All participants will also have a bronchoscopy and provide sputum, saliva, and buccal smear samples at 12 months. If you have been treated for HNSCC, you will have a laryngoscopy at 12 months.

After the first year, you will be followed for a minimum of 2 more years and a maximum of 6 years. You will have physical exams at 24 and 36 months. You will have blood draws (about 3 teaspoons for routine tests and 4 teaspoons for research purposes), a chest x-ray and a chest CT at 18, 24, 30 and 36 months. After 36 months, you will have a physical exam by a physician or nurse every 6 months for up to 6 years. Every 12 months the physical exam will be done by a physician. The other physical exams will be done by a nurse. You will have blood drawn for routine tests (about 3 teaspoons) and research purposes (about 4 teaspoons) every 12 months.

This research study includes two bronchoscopies done one year apart. These bronchoscopies are being done primarily for research purposes and are unlikely to provide information useful in your individual treatment. These bronchoscopies do have risks associated with them. These risks are described in section 4 of this informed consent document.

Recent research on early stage NSCLC indicates that adjuvant chemotherapy after surgery increases the length of time a person may survive and the length of time before cancer recurs. However, this adjuvant chemotherapy also has side effects that can be severe and in rare cases fatal. If you have had surgery for NSCLC and wish to receive adjuvant chemotherapy, you may only enroll in this study and Protocol 2003-0424 after you have completed the adjuvant chemotherapy.

As part of this study you will provide samples of your lung tissue, saliva, blood, and scrapings from the inside of your cheek. Fluid and mucous collected during the bronchoscopies will also collected. These samples will be studied by scientists to learn about genes and proteins in people who have been treated for early NSCLC or HNSCC. The samples will also be used to grow cells and cultures that will be used to test chemotherapy drugs. These cells and cultures will also be used to learn about genes and proteins.

This is an investigational study. Celecoxib is a commonly used drug that is approved by the FDA for treatment of arthritis, colon polyps, and pain. The use of celecoxib to help prevent cancer is approved by the FDA for research only. A total of up to 70 individuals will take part in this multicenter study. Up to 50 will be enrolled at UT MD Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with either: a) histologically proven stage I, II, or IIIa NSCLC who have undergone a complete surgical resection of the primary tumor OR b) stage I or II HNSCC who have undergone definitive local treatment (surgery or radiation therapy).
2. HNSCC patients: Definitive local treatment </= 12 months prior to trial enrollment. NSCLC patients: Surgery </= 12 months prior to trial enrollment.
3. No evidence residual cancer
4. Smoking history of at least 10 pack years. May be current or former smoker.
5. Performance status of < = 2 (Zubrod)
6. Age =>18 years
7. Participants must have no contraindications for undergoing bronchoscopy.
8. Patients must have no active pulmonary infections.
9. Participants must not be taking oral non-steroidal anti-inflammatory drugs on a regular basis.
10. Participants must have the following blood levels: total granulocyte count >1500; platelet count > 100,000; total bilirubin < = 1.5 mg. %; and creatinine < = 1.5 mg %.
11. Participants must complete the pretreatment evaluation and must consent to bronchoscopy and to endobronchial biopsy for biomarker studies.
12. All subjects who agree to participate will be given a written and verbal explanation of the study requirements and a consent form that must be signed prior to registration. Subjects will be informed that (a) they must be willing to take capsules daily for the duration of the trial, (b) they must be willing to take biopsies through bronchoscopy and give blood samples at the specified times, (c) they must schedule and keep the specified follow-up visits with their physicians and the study clinics, and (d) side effects and health risks may occur, as described in the informed consent form.
13. Participant must be enrolled in UT MD Anderson Cancer Center protocol #2003-0424 titled "A Phase IIb Vanguard Study Characterizing the Occurrence of Recurrent or Second Primary Tumors in Patients with a Prior History of a Definitively Treated Stage I/II Head and Neck or Non-Small Cell Cancer who are Current or Former Smokers."
14. Patients with prior head and neck cancer only: Participants must have no contraindications for undergoing laryngoscopy.
15. Subject must be considered legally capable of providing his or her own consent for participation in this trial.

Exclusion Criteria:

1. History of radiation therapy to the chest. For those patients with head and neck cancer who received radiation, no more than 10% of the lung volume (apices) may be included.
2. History of systemic chemotherapy. Exception: NSCLC patients may have had up to 4 cycles of platinum-based doublet therapy.
3. Pregnant or breast-feeding (a negative pregnancy test within 72 hours of enrollment for women with child-bearing potential is required)
4. Participants with active gastric or duodenal ulcers or a history of ulcers requiring prophylactic H2 blockers.
5. Participants with active pulmonary infections or recent history of pulmonary infection (within one month).
6. Participants with acute intercurrent illness
7. Participants requiring chronic ongoing treatment with Nonsteroidal anti-inflammatory drugs (NSAIDs). (Casual or non-prescribed use of NSAIDs is permitted as long as their use does not exceed one week at a time.)
8. Participants who are allergic to aspirin or sulfanamides.
9. Patients may not take high dose antioxidants (vitamins E or C) during the study period. "High dose" will be determined by the study investigators.
10. Patients may not take high dose synthetic or natural Vitamin A derivatives (> 10,000 IU per day).
11. History of biologic therapy
12. Women of childbearing potential and men with partners of childbearing potential who are not using an effective method of contraception. Use of contraception will be verified at office visits during first year on study.
13. History of cardiovascular diseases that might include one of the following: myocardial infarction, angina, coronary angioplasty, congestive heart failure, stroke, or coronary bypass surgery.
14. Diagnosis of diabetes
15. History of deep venous thrombosis, pulmonary embolism, systemic lupus erythematosus, family history of protein S or C deficiencies, prior heparin-induced thrombocytopenia, or known Factor V Leiden mutation.
16. Family history of premature CAD. This is defined as individuals with either: 1) father with MI prior to age 55, or 2) mother with MI prior to age 60.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2005-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Waun K. Hong, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: September 29, 2005 to December 18, 2007. Patients were recruited at UT MD Anderson Cancer Center.
Pre-assignment Details: One patient registered determined to be inevaluable. Trial termination due to poor accrual and study program redesign.
Groups:
- Celecoxib Treatment: Celecoxib 600 mg orally daily
Period: Overall Study
Arm/Group | Celecoxib Treatment | No Treatment
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Celecoxib Treatment | No Treatment | Total
Number analyzed (Participants) | 1 | 0 | 1
Age Categorical [Number; unit: years]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 0 |  | 0
Gender [Number; unit: participants]
  Female | 1 |  | 1
  Male | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Histological Responses
Description: Number of patients with histological response based on changes in bronchoscopies from baseline to 12 months.
Time Frame: Baseline to 12 months
Population: No analysis. One registered patient inevaluable for response, study terminated early.
Arm/Group | Celecoxib Treatment | No Treatment
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 21 months
Arm/Group | Celecoxib Treatment | No Treatment
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes